CLINICAL TRIAL: NCT06893822
Title: The Effect of Griffonia Simplicifolia on Pain Intensity, Central and Peripheral Sensitization, Painmodulation in Healthy Volunteers - A Randomized, Double-blinded, Placebo-controlled, Cross-over Study
Brief Title: The Effect of Griffonia Simplicifolia on Pain Intensity, Central and Peripheral Sensitization, Painmodulation in Healthy Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1308/2024
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Central Sensitisation; Peripheral Sensitization; Neuroinflammatory Response
Keywords: Griffonia simplicifolia; 5-HTP; Peripheral Sensitisation; Central Sensitisation
MeSH Terms: conditions — Chronic Pain | interventions — Griffonia simplicifolia lectins

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Griffonia simplicifolia) - Placebo (Experimental): Participants receive Griffonia s. 1x day for 28 days, 4 weeks wash out will follow, then they receive placebo for 28 days.
  Interventions: Dietary Supplement: Griffonia simplicifolia; Other: Placebo
- Placebo - Verum (Griffonia simplicifolia) (Placebo Comparator): Participants receive placebo 1xd ay for 28 days, 4 weeks washout will follow, then they receive Griffonia s. for 28 days
  Interventions: Dietary Supplement: Griffonia simplicifolia; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Griffonia simplicifolia — Griffonia simplicifolia 1x/day
Other: Placebo — Placebo 1x/day

SUMMARY:
This planned study is based on a randomized, placebo-controlled cross-over design.

Griffonia simplicifolia contains the serotonin-precursor 5-hydroxytryptophan (5-HTP), an endogenous amino acid. 5-HTP can cross the blood-brain barrier and is converted to serotonin. Low serotonin levels are associated with depression, anxiety disorders and sleep disorders, among others. Griffonia simplicifolia is marketed as a food supplement in accordance with EU Directive 2002/46/EC. Several clinical studies have examined the efficacy of 5-HTP in chronic pain conditions.

The data suggest a clinical analgesic efficacy, without, however, allowing conclusions about the underlying mechanisms. These have not yet been investigated in a human experimental pain model. The aim of the study is to investigate the influence of 5-HTP in peripheral and central sensitization, as well as descending inhibitory pathways by Quantitative Sensory Testing (QST). These findings are of great relevance for a better understanding of clinical efficacy.

For this purpose, "repetitive phasic heat application" is a validated method for achieving short-term peripheral and central sensitization. As a non-invasive human pain model, it is therefore well suited for investigating the analgesic and anti-hyperalgesic effects of drugs.

Furthermore, the influence of Griffonia simplicifolia on mood (depression, anxiety), memory, sleep quality and psychological well-being will be investigated by using psychological questionnaires as secondary target variables.

DETAILED DESCRIPTION:
Griffonia simplicifolia contains the serotonin-precursor 5-hydroxytryptophan (5-HTP), an endogenous amino acid. 5-HTP can cross the blood-brain barrier and is converted to serotonin. Low serotonin levels are associated with depression, anxiety disorders and sleep disorders, among others. Griffonia simplicifolia is marketed as a food supplement in accordance with EU Directive 2002/46/EC. Several clinical studies have examined the efficacy of 5-HTP in chronic pain conditions.

The data suggest a clinical analgesic efficacy, without, however, allowing conclusions about the underlying mechanisms. These have not yet been investigated in a human experimental pain model. The aim of the study is to investigate the influence of 5-HTP in peripheral and central sensitization, as well as descending inhibitory pathways by Quantitative Sensory Testing (QST). These findings are of great relevance for a better understanding of clinical efficacy.

An effect on peripheral sensitization speaks in favor of use in acute somatic pain. However, if the effect can be explained by central mechanisms, its use would be recommended in chronic or neuropathic pain. For this purpose, "repetitive phasic heat application" is a validated method for achieving short-term peripheral and central sensitization. As a non-invasive human pain model, it is therefore well suited for investigating the analgesic and anti-hyperalgesic effects of drugs.

Furthermore, the influence of Griffonia simplicifolia on mood (depression, anxiety), memory, sleep quality and psychological well-being will be investigated by using psychological questionnaires as secondary target variables.

The following questions were be answered in this study:

* Can the administration of Griffonia simplicifolia reduce spontaneous pain following repetitive phasic heat application?
* Does the intake of Griffonia simplicifolia modulate central sensitization?
* Does the intake of Griffonia simplicifolia influence peripheral sensitization?
* Can the descending inhibitory pathways be modulated through the administration of Griffonia simplicifolia?
* Can the intake of Griffonia simplicifolia enhance memory performance?
* Is a reduction in depression scores achievable through Griffonia simplicifolia administration?
* Can anxiety scores be reduced by the administration of Griffonia simplicifolia?
* Is sleep quality improved with the intake of Griffonia simplicifolia?

The following methods were used to answer these questions:

* Spontaneous pain was determined using the numeric rating scale (NRS).
* Central sensitization was evaluated by pain sensitivity to mechanical stimuli, i.e. pinprick hyperalgesia or allodynia.
* An effect on peripheral sensitization was investigated by measuring the heat detection threshold and heat pain threshold.
* The body's own pain inhibition was evaluated by means of a "conditioned pain modulation" test.
* The influence on mood (depression and anxiety), sleep, memory and well-being were evaluated using psychological survey instruments.

Null hypothesis:

The intake of Griffonia simplicifolia 1 x 100 mg over 28 days does not change the spontaneous pain after repetitive phasic heat application compared to placebo intake.

Alternative hypothesis:

The intake of Griffonia simplicifolia 1x 100 mg over 28 days changes the spontaneous pain after repetitive phasic heat application compared to placebo intake.

Secondary hypotheses:

* There is a significant difference in the size of the mechanical allodynia distance and the flare area after repetitive phasic heat application when taking Griffonia simplicifolia compared to placebo.
* There is a change in pinprick hyperalgesia with Griffonia simplicifolia compared to placebo after repetitive phasic heat application.
* The intake of Griffonia simplicifolia leads to a change in the heat perception and pain threshold compared to placebo intake after repetitive phasic heat application.
* The intake of Griffonia simplicifolia leads to a change in "conditioned pain modulation" compared to placebo intake.

Study design:

This study is based on a randomized, double-blind, placebo-controlled, cross-over design.

After recruitment, information and inclusion of the study participants, the first baseline measurement consisting of the sensory parameters and psychological questionnaires is carried out. The test subjects are randomized into two groups. They take either the test substance (verum; 100 mg Griffonia simplicifolia daily) or the placebo for 28 days. Both the participants and the study staff responsible for collecting the measurement parameters are blinded to the order in which the tablets are taken.

After recruitment, information and inclusion of the subjects in the study, the first baseline measurement is performed. After 28 days, during which either the verum or study substance is taken, the influence on the "conditioned pain modulation" is measured. The repetitive phasic heat application according to the published procedures follows. A 3x3cm area on the volar forearm is heated repeatedly using a TSA-II NeuroSensoryAnalyser. The thermode starts at 32.0°C and heats up to 48.0°C at 10°C/sec and cools down to 32.0°C after 6 seconds. This is repeated 6 times in total. This is followed by a 30 second pause and then 6 more heatings. A total of 10 blocks with 6 heatings each are performed.

At the end of the last block, spontaneous pain is determined using the Visual Analogue Scale.

Since primary and secondary hyperalgesia is most pronounced at 1 hour after repetitive phasic heat application, 60 minutes after the last heating, the measurement of allodynia distance and pinprick hyperalgesia is performed in immediate temporal sequence and the heat pain and perception threshold is determined.

After a 4-week wash-out phase, the third study visit is held. It included again the baseline measurement. Subsequently, the other substance is taken for 28 days. This is followed by the fourth study visit including the survey of the sensory parameters and the repetitive phasic heat application.

To investigate the influence of Griffonia simplicifolia on the psyche, the participants answered various psychological questionnaires during all four study visits. These focused on depression, anxiety, sleep quality, well-being, memory and medication adherence.

Sample size calculation:

The study by Jurgens et al., in which repetitive phasic heat application was tested in healthy subjects, was used as the data basis (Jürgens TP, Sawatzki A, Henrich F, Magerl W, May A. An improved model of heat-induced hyperalgesia--repetitive phasic heat pain causing primary hyperalgesia to heat and secondary hyperalgesia to pinprick and light touch. PLoS One. 2014 Jun 9;9(6):e99507).

In this publication, the mean value for maximum pain was 72.2 (numerical scale 0-100), the standard deviation was given as 5.4. If the base data for the case number calculation are taken more conservatively and doubled (SD = 10.8), a sample size of 20 would have a power of 0.93 to detect a difference of 10 units on a 0-100 numerical pain scale using a paired samples t-test with alpha = 0.05 and drop-out rate of 0.2.

Statistics:

No data are available on the probability of a period effect. The probability of a carryover effect is low, as the washout interval of 28 days was chosen to be sufficiently long, as a HWZ of 5-HTP of approx. 4 h is assumed.

After completion of the data collection, descriptive statistics were performed (separately for treatment A and B as well as period 1 and 2). Continuous values were summarized using mean, median, standard deviation, minimum and maximum. The Shapiro-Wilk test is used to verify a possible normal distribution. This is followed by a comparison of the results of both periods and treatment series (AB vs. BA) as well as a check for a carryover effect (comparison of the first periods of treatments A and B using an unpaired t-test). The further statistical procedure depends, among other things, on the existence of a carryover effect and the completeness of the data. Accordingly, if the preconditions are met, either a linear mixed model (LMM; e.g. for missing values or dropouts) or an ANOVA (advantageous when considering period and subject effects) is used. If there is no normal distribution, a Wilcoxon signed rank test can be used. With a p-value <0.05, the null hypothesis was rejected. Qualitative data is evaluated using a chi-square test. The effect size is calculated by dividing the Z value by the square root of N.

Study substance:

The participants each receive 28 capsules containing either Griffonia simplicifolia 100 mg (Nutricost) or an optically identical placebo (veggie capsules, size 1, maltodextrin filler) manufactured in a pharmacy. It is taken at 24-hour intervals. The last dose is taken in the morning before the study visit. To increase adherence to therapy, an electronic reminder will be sent via cell phone. Capsules that have not been taken should be brought to the study visit after the respective intake interval.

Parameter:

Spontaneous pain:

Directly after the last heat application, the spontaneous pain is recorded using the VAS scale, which is used throughout the LKH Univ.-Klinikum Graz.

Allodynia:

Starting from the center of the thermal application, a von Frey filament (128 mN) is applied to the skin in 4 radial lines at a 5 mm interval, first from the inside to the outside, then from the outside to the inside, and the distance at which an unpleasant pointed sensation first occurs is determined. The 8 measurements are averaged.

Pinprick hyperalgesia:

By means of a pinprick with 256 mN a pointed stimulus is applied. The test site is 5 cm proximal to the center of the thermal stimulation area. A numerical scale (0-100) is used to measure how painful this stimulus is.

Heat pain and perception threshold:

The heat detection threshold and the heat pain threshold are determined according to the guidelines of the German Research Association for Neuropathic Pain, which involves heating the skin with TSA-II NeuroSensoryAnalyser. The test person can stop the heating by pressing a stop button. This should be done at the first time he/she notices that the skin is warming up (heat detection threshold) or at the time he/she notices a pulling, burning or pricking sensation in addition to the feeling of heat (heat pain threshold). The measurements are taken 3 times each and the results are averaged.

Conditioned pain modulation:

Conditioned pain modulation describes the function of the descending, pain-inhibiting system. First, the force with which pressure on the adductor pollicis brevis muscle of the non-dominant hand is not only perceived as pressure, but also as a stabbing, burning or pulling sensation is determined using a pressure gauge. Subsequently, the contralateral hand is immersed in ice water until the subject feels a pain intensity of NRS 40 (101-part scale). The pressure pain threshold is then immediately raised again.

The following psychological questionnaires were answered at the four study visits:

Beck's Depression Inventory (BDI-II), Beck's Anxiety Inventory (BAI), Pittsburgh Sleep Quality Index (PSQI), WHO-5 questionnaire, Modul "Memory" of the Neuropsychological Assessment Battery (NAB) and Medication Adherence Report Scale (MARS-d; only at the 2nd and 4th study visit).

Adverse effects:

Possible adverse effects are assessed and documented at each study visit. In addition, the subjects are informed about the necessity of immediate telephone contact in case of the occurrence of undesirable side effects.

Recruitment and informed consent:

Recruitment of participants is done by posting on notice boards at the ÖH an der Med-Uni Graz (main building) and the outpatient pain clinic

Participants are asked orally whether they participate in another study at the same time or whether a required period of time has elapsed since participation in another study. They confirm this with their signature.

A physician involved in the study will provide the information. Consent is then given by signing a written information sheet.

The investigation of pain and perception thresholds according to the specifications of the "German Research Association for Neuropathic Pain" is an established procedure in both human research and clinical investigation. No danger is to be expected for the individual test person.

The application of "repetitive phasic heat application" is an established human pain model. The maximum heat exposure of 48°C does not lead to skin damage. The changes in pain sensitivity are locally very limited and normalize within a few hours.

If the individual test person is willing to be exposed to a pain stimulus for a limited period of time, there is no foreseeable risk for him/her.

Griffonia simplicifolia is marketed as a food supplement in accordance with EU Directive 2002/46/EC.

Possible side effects are dizziness, headaches, photosensitivity and sedation due to the central effect. Nausea, vomiting, diarrhea, bloating or stomach pain may also occur.

Contraindications include severe hepatic and renal insufficiency. Due to a lack of studies, it is not recommended for use during pregnancy and breastfeeding.

Taking high doses of Griffonia simplicifolia or the main ingredient 5-hydroxytryptophan (5-HTP) together with antidepressants (such as SSRIs), MAO inhibitors or St. John's wort may result in a risk of interaction in the form of serotonin syndrome.

In the past, so-called eosinophilia-myalgia syndrome (EMS) has occurred after taking individual tryptophan-containing products. EMS can lead to severe muscle pain, skin changes, cramps, fever and damage to the heart and lungs.

5-HTP is closely related to the natural amino acid tryptophan, which is why its influence on the possible development of EMS is also being discussed. However, as the connection could not be conclusively proven, tryptophan and 5-HTP are still available. The clinical picture did not occur in the existing studies either. Statistical studies on a larger patient collective are lacking.

ELIGIBILITY:
Exclusion Criteria:

* pregnancy or breastfeeding.
* renal or hepatic insufficiency
* neurological/dermatological/cardiovascular diseases
* chronic pain and/or use of analgesics
* intake of antidepressants
* intake of MAO inhibitors
* intake of sleep medication
* intake of St. John's wort
* allergy to Griffonia simplicifolia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-12 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in spontaneous pain intensity | -->Day 0 -->Day 28 before repeated heat application --> Day 28 1 hour after repeated heat application --> Day 56 -->Day 84 before repeated heat application -->Day 84 1 hour after repeated heat application
  is measured on a visual analogue scale (0 means no pain and 10 means the worst imaginable pain)

SECONDARY OUTCOMES:
Change in Allodynia | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 84 before repeated heat application -->Day 84 1 hour after repeated heat application
  measured in radial distance in mm
Change in Hyperalgesia | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 84 before repeated heat application -->Day 84 1 hour after repeated heat application
  measured with pinpricks, that are preset different peak stimulus. A numerical scale (0-100) is used to measure how painful the stimulus is.
Change in heat detection threshold | ->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 84 before repeated heat application -->Day 84 1 hour after repeated heat application
  measured in degrees C°
Change in heat pain threshold | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 --> Day 84 before repeated heat application -->Day 84 1 hour after repeated heat application
  measured in degrees C°
Change in conditioned pain modulation | Time Frame: -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 84 before repeated heat application -->Day 84 1 hour after repeated heat application
  measures the descending analgesic System with the help of a pressure algometer in kg
Psychological Questionnaires | All four study visits: BDI-II, BAI, PSQI, WHO-5 questionnaire, Modul "Memory" of the Neuropsychological Assessment Battery (NAB); Only at the 2nd and 4th study visit: Medication Adherence Report Scale (MARS-d).
  The participants answered psychological questionnaires on depression, anxiety, sleep quality, well-being, memory and medication adherence.
  The questionnaires were always handed out before the sensory tests.
  The following psychological questionnaires were answered at the four study visits:
  Depression: Beck's Depression Inventory (BDI-II) Anxiety: Beck's Anxiety Inventory (BAI) Sleep quality: Pittsburgh Sleep Quality Index (PSQI) Well-being: WHO-5 questionnaire Memory: Modul "Memory" of the Neuropsychological Assessment Battery (NAB) Medication adherence (only at the 2nd and 4th study visit): Medication Adherence Report Scale (MARS-d)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No